CLINICAL TRIAL: NCT03454412
Title: A Pilot Study of Hand Function in Children With Cerebral Palsy Undergoing Intensive Neurophysiological Rehabilitation
Status: Completed | Type: Observational
Sponsor: International Clinic of Rehabilitation, Ukraine (Other)
Responsible Party: Principal Investigator, Oleh Kachmar, Head of Innovative Technologies Department, International Clinic of Rehabilitation, Ukraine
Other Study IDs: N-02-2018
Record Dates: First submitted 2018-02-27; First posted 2018-03-05 (Actual); Results first posted 2021-05-25 (Actual); Last update posted 2021-05-25 (Actual); Status verified 2021-04

CONDITIONS: Cerebral Palsy
Keywords: Cerebral Palsy; Rehabilitation; Hand
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Intensive Neurophysiological Rehabilitation — Intensive Neurophysiological Rehabilitation System (INRS) is a combination of different treatment modalities that complement and reinforce each other. It includes spinal manipulative therapy, physical therapy, occupational therapy, joints mobilization techniques, special massage therapy, mechanotherapy, computer games therapy and other treatments with daily duration up to 4 hours.

SUMMARY:
The aim of the study is to observe the effects of Intensive Neurophysiological Rehabilitation System on hand function in children with spastic cerebral palsy.

DETAILED DESCRIPTION:
Intensive Neurophysiological Rehabilitation System is a novel multimodal rehabilitation approach that combines different treatment modalities. The treatment course lasts for 2 weeks with daily therapy up to 4 hours. Main treatment programs include biomechanical correction of the spine, extremity joint mobilization, physical and occupational therapy, reflexotherapy, special massage system, rhythmical group exercises, mechanotherapy and computer games therapy and some other.

Preliminary observational studies indicate an improvement of gross and fine motor functions in children with Cerebral Palsy after the treatment course.

The aim of the study is to observe the effects of Intensive Neurophysiological Rehabilitation System on hand function in children with spastic cerebral palsy.

About 50 patients with spastic forms of cerebral palsy with mild to moderate impairment of hand function (Level I to III according to Manual Abilities Classification System) would be evaluated before and after the two-week treatment course.

This study may help to generate the hypothesis of the effects of the Intensive treatment course on hand function abilities and to prepare a future randomized controlled trial.

ELIGIBILITY:
Inclusion Criteria:

* Spastic cerebral palsy: uni- and bilateral
* Age: 6-15
* Level I-III according to Manual Ability Classification System (MACS)

Exclusion Criteria:

* Ataxic or dyskinetic cerebral palsy
* Non-cooperative behavior
* Moderate to severe mental deficit
* Severe contractures of upper extremity joints
* Upper extremities trauma within 6 months prior to the study
* Previous hand surgery
* Epilepsy with frequent seizures

Ages: 6 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children with spastic cerebral palsy aged six to fifteen undergoing Intensive Neurophysiological Rehabilitation.
Sampling Method: Non-Probability Sample
Enrollment: 44 (Actual)
Dates: Start 2018-03-19 (Actual); Primary Completion 2019-05-01 (Actual); Study Completion 2019-05-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Oleh Kachmar, MD, PhD, Principal Investigator — International Clinic of Rehabilitation, Ukraine
Locations (1):
- International Clinic of Rehabilitation, Truskavets, Lviv Oblast, Ukraine

IPD SHARING:
Plan to Share IPD: No
No individual participants data will be shared.

REFERENCES:
- [Background] Kachmar O, Voloshyn T, Hordiyevych M. Changes in Muscle Spasticity in Patients With Cerebral Palsy After Spinal Manipulation: Case Series. J Chiropr Med. 2016 Dec;15(4):299-304. doi: 10.1016/j.jcm.2016.07.003. Epub 2016 Sep 28. PMID 27857638
- [Background] Koziavkin VI, Voloshin TB, Gordievich MS, Kachmar OA. [Changes of motor function in patients with cerebral palsy during the treatment using the intensive neurophysiological rehabilitation system]. Zh Nevrol Psikhiatr Im S S Korsakova. 2012;112(7 Pt 2):14-7. Russian. PMID 23330186
- [Background] Kozyavkin VI, Kachmar OO. Rehabilitation outcome assessment methods in Intensive neurophysiological rehabilitation system. Ukrayinskyj Medychnyj Chasopys. 2003;3(35):61-66. [in Ukrainian]
- [Background] Kozyavkin VI, Babadagly MO, Lun GP. : . Intensive Neurophysiological Rehabilitation System-the Kozyavkin Method. A Manual for Rehabilitation Specialists, Design studio Papuga; Lviv, Ukraine, 2012

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients that met inclusion criteria and scheduled for the treatment to the International Clinic of Rehabilitation were invited.
Pre-assignment Details: 32 of total enrolled 44 participants met inclusion criteria and were included into the study
Groups:
- Intensive Neurophysiological Rehabilitation: Patients undergoing 2 weeks treatment course
Period: Baseline Assesment
Arm/Group | Intensive Neurophysiological Rehabilitation
Started | 44
Completed | 32
Not Completed | 12
Not completed — Physician Decision | 12
Period: Treatment Course
Arm/Group | Intensive Neurophysiological Rehabilitation
Started | 32
Completed | 32
Not Completed | 0
Period: Final Assesment
Arm/Group | Intensive Neurophysiological Rehabilitation
Started | 32
Completed | 32
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Intensive Neurophysiological Rehabilitation: Patients undergoing two-weeks treatment course of Intensive Neurophysiological Rehabilitation
Arm/Group | Intensive Neurophysiological Rehabilitation
Number analyzed (Participants) | 32
Age, Continuous [Mean (Standard Deviation); unit: years] | 10.2 (2.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 18
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 32
  More than one race | 0
  Unknown or Not Reported | 0
Dominant hand [Count of Participants; unit: Participants]
  Right hand dominant | 18
  Left hand dominant | 14
Diagnosis [Count of Participants; unit: Participants]
  Cerebral Palsy, spastic diplegia | 11
  Cerebral Palsy, spastic quadriplegia | 21
Manual Ability Classification System level [Count of Participants; unit: Participants] — The Manual Ability Classification System (MACS) describes how children with cerebral palsy use their hands to handle objects in daily activities. MACS includes five levels.
  Level I - Handles objects easily and successfully. Level II. Handles most objects but with somewhat reduced quality /speed. Level III - Handles objects with difficulty; needs help to prepare and/or modify activities. Level IV. Handles a limited selection of easily managed objects in adapted situations. Level V. Does not handle objects and has severely limited ability to perform even simple actions.
  Participants
    Level I | 7
    Level II | 15
    Level III | 10
GMFCS level [Count of Participants; unit: Participants] — The Gross Motor Function Classification System or GMFCS is a 5 level clinical classification system that describes the gross motor function of people with cerebral palsy on the basis of self-initiated movement abilities Level I - Walks without Limitations Level II - Walks with Limitations Level III - Walks Using a Hand-Held Mobility Device Level IV - Self-Mobility with Limitations; May Use Powered Mobility Level V - Transported in a Manual Wheelchair
  Participants
    GMFCS Level I | 8
    GMFCS Level II | 10
    GMFCS Level III | 13
    GMFCS Level IV | 1

OUTCOME MEASURES:

1. Primary Outcome: Jebsen Taylor Hand Function Test for Dominant Hand
Description: The Jebsen Hand Function Test for Dominant Hand assesses hand function activities during performance of activities of daily living of the dominant hand.
  Test quantifies the time it takes for the subject to do the following standardized functional tasks with one hand: turning over cards, picking up small items, simulating feeding, stacking checkers, picking up light cans, and picking up heavy cans.Total score is the sum of time taken for each sub-test, which are rounded to the nearest second. Shorter times indicate better performance.
Time Frame: Baseline and post intervention (after the two-week treatment course)
Measure: Mean (Standard Deviation); unit: seconds
Groups:
- Intensive Neurophysiological Rehabilitation: Patients undergoing two-week treatment course of Intensive Neurophysiological Rehabilitation
Arm/Group | Intensive Neurophysiological Rehabilitation
Number analyzed (Participants) | 32
seconds
  Baseline | 130.1 (83)
  Post intervention | 115.2 (77)

2. Primary Outcome: Jebsen Taylor Hand Function Test for Non-Dominant Hand
Description: The Jebsen Hand Function Test for Non-Dominant Hand assesses hand function activities during performance of activities of daily living of the non-dominant hand.
  Test quantifies the time it takes for the subject to do the following standardized functional tasks with one hand: turning over cards, picking up small items, simulating feeding, stacking checkers, picking up light cans, and picking up heavy cans.Total score is the sum of time taken for each sub-test, which are rounded to the nearest second. Shorter times indicate better performance.
Time Frame: Baseline and post intervention (after the two-week treatment course)
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Intensive Neurophysiological Rehabilitation
Number analyzed (Participants) | 32
seconds
  Baseline | 191.5 (109)
  Post intervention | 181.4 (114)

3. Secondary Outcome: ABILHAND-Kids Test Score
Description: Ability of the hand (ABILHAND)-Kids is a measure of manual ability for children with upper limb impairments. The scale measures a person's ability to manage daily activities that require the use of the upper limbs. The Parent is asked to fill in the questionnaire by estimating their child's performance of 21 manual activities on a 3-level scale (impossible, difficult, easy).
  Measured score is expressed in logits ranging from "- 7" to "+7". The logit is a linear unit that expresses the odds of success of the patient on any given item. The higher score indicates better function.
Time Frame: Baseline and post intervention (after the two-week treatment course)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intensive Neurophysiological Rehabilitation
Number analyzed (Participants) | 32
score on a scale
  Baseline | 1.92 (1.8)
  Post intervention | 2.26 (2.0)

4. Secondary Outcome: Box and Blocks Test for Dominant Hand
Description: The test is measuring the dexterity of the dominant hand. The score is the number of blocks carried by the dominant hand from one compartment to the other in one minute.
Time Frame: Baseline and post intervention (after the two-week treatment course)
Measure: Mean (Standard Deviation); unit: blocks carried
Arm/Group | Intensive Neurophysiological Rehabilitation
Number analyzed (Participants) | 32
blocks carried
  Baseline | 33.5 (12)
  Post intervention | 35.5 (13)

5. Secondary Outcome: Box and Blocks Test for Non-Dominant Hand
Description: The test is measuring the dexterity of the non-dominant hand. The score is the number of blocks carried by the non-dominant hand from one compartment to the other in one minute.
Time Frame: Baseline and post intervention (after the two-week treatment course)
Measure: Mean (Standard Deviation); unit: blocks carried
Arm/Group | Intensive Neurophysiological Rehabilitation
Number analyzed (Participants) | 32
blocks carried
  Baseline | 28.0 (11)
  Post intervention | 29.8 (11)

6. Secondary Outcome: Maximum Grip Force of the Dominant Hand
Description: Grip force of the Dominant Hand is measured by Jamar hand dynamometer in kilograms. All children had three trials and the best result was recorded
Time Frame: Baseline and post intervention (after the two-week treatment course)
Measure: Mean (Standard Deviation); unit: kilogram
Arm/Group | Intensive Neurophysiological Rehabilitation
Number analyzed (Participants) | 32
kilogram
  Baseline | 12.1 (5.6)
  Post intervention | 11.8 (5.4)

7. Secondary Outcome: Maximum Grip Force of the Non-Dominant Hand
Description: Grip force of the Non0Dominant Hand is measured by Jamar hand dynamometer in kilograms. All children had three trials and the best result was recorded
Time Frame: Baseline and post intervention (after the two-week treatment course)
Measure: Mean (Standard Deviation); unit: kilogram
Arm/Group | Intensive Neurophysiological Rehabilitation
Number analyzed (Participants) | 32
kilogram
  Baseline | 10.8 (6.0)
  Post intervention | 10.5 (4.9)

ADVERSE EVENTS:
Time Frame: Two weeks - from Baseline assesment till the Post intervention assesment
Description: Default
Arm/Group | Intensive Neurophysiological Rehabilitation
All-Cause Mortality (participants affected / at risk) | 0/32
Serious Adverse Events (participants affected / at risk) | 0/32
Other Adverse Events (participants affected / at risk) | 0/32

LIMITATIONS AND CAVEATS:
Short-term period of study, lack of blinding due to the pre-post design with the absence of the control group, and relatively small sample size.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2017-05-15): https://cdn.clinicaltrials.gov/large-docs/12/NCT03454412/Prot_SAP_ICF_000.pdf